CLINICAL TRIAL: NCT05895786
Title: A PHASE 3, MULTICENTER, DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED STUDY TO EVALUATE THE EFFICACY AND SAFETY OF PF-06823859 IN PARTICIPANTS WITH ACTIVE IDIOPATHIC INFLAMMATORY MYOPATHIES (INCLUDING PARTICIPANTS WITH ACTIVE DERMATOMYOSITIS OR POLYMYOSITIS)
Brief Title: A Study to Understand How the Study Medicine (PF-06823859) Works in People With Active Idiopathic Inflammatory Myopathies [Dermatomyositis (DM) and Polymyositis (PM)]
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C0251006; 2022-502739-20-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-04-27; First posted 2023-06-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Myositis
Keywords: Dermatomyositis; Polymyositis
MeSH Terms: conditions — Myositis; Dermatomyositis; Polymyositis

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group study to assess whether the study medicine will work to lessen muscle weakness and skin symptoms in adults with active polymyositis (PM) or dermatomyositis (DM). Eligible participants are required to have active disease at the time of enrollment and are required to enter the study on protocol-permitted standard of care (SOC) background medication.
  The study will be conducted in 2 parallel cohorts: Cohort 1 (DM) and Cohort 2 (PM).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The sponsor, participants, and site personnel (including the investigator) will be masked to study treatment and will not know whether active study medication or placebo is being administered to participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-06823859 (Experimental): Participants will receive PF-06823859 via intravenous infusion every 4 weeks.
  Interventions: Drug: PF-06823859
- Placebo (Placebo Comparator): Participants will receive placebo via intravenous infusion every 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06823859 — anti-interferon beta therapy
  Arms: PF-06823859
Drug: Placebo — Placebo for PF-06823859
  Arms: Placebo

SUMMARY:
The purpose of the study is to understand how the study medicine PF-06823859 (dazukibart) works in people with idiopathic inflammatory myopathies (DM and PM). These disorders cause inflammation that weakens the muscles that are important for movement and may also cause skin rash in people with DM.

This study is seeking participants who:

* Are 18 years of age or older or minimum legal adult age as defined per local regulation, whichever is greater
* Have active DM or active PM.
* Are receiving a stable dose of 1 corticosteroid taken by mouth and/or 1 traditional immunosuppressant.

  * Note: Corticosteroids and immunosuppressants are medicines that help reduce inflammation and may signal to the immune system not to attack the body.

Dermatomyositis (DM) is a rare disease that causes muscle inflammation that results in muscle weakness and low muscle stamina. Patients with DM have a characteristic skin rash. Polymyositis (PM) is a rare disease that involves mainly muscle inflammation resulting in muscle weakness, that can sometimes be painful. Patients with DM and PM may have trouble going up the steps, walking or getting to a standing position.

Some of the participants will receive the study medicine (dazukibart) and some will receive placebo (which is similar to study medicine but contains no medicine in it).

The study medicine or placebo will be given as an intravenous (IV) infusion (directly into the veins), which takes about 1 hour; every 4 weeks from Day 1 to Week 48 of the study. Both dazukibart and placebo and will be given at the study site.

The study will compare the experiences of people receiving study medication to those of the people who do not. This will help to see if dazukibart is safe and effective.

Participants will take part in this study for about 13 months. During this time, participants will have 15 study visits. These visits will be performed at the study site.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults (≥18 years old or minimum legal adult age as defined per local regulation, whichever is greater)
* Active dermatomyositis (DM) or polymyositis (PM) with age of onset

  * 18 years old.
* Must be receiving a stable dose of standard of care (SOC) background medications at the time of enrollment.

Exclusion Criteria:

* Myositis due to non-Idiopathic inflammatory myopathies (non-IIM)
* Existing diagnosis of inclusion body myositis (IBM)
* Presence of immune-mediated necrotizing myositis (IMNM)
* Myositis with end-stage organ involvement
* Active bacterial, viral or fungal infections or hospitalizations for serious infections within 60 days prior to enrollment
* History of recurrent bacterial, viral, fungal, mycobacterial or other infections
* Clinically significant finding on a chest x-ray
* Have cancer or a history of cancer within 5 years of screening
* Significant current or prior disease conditions that may interfere with the response to or safety of the study medicine, including but not limited to:
* history of major organ transplant
* acute coronary syndrome or any history of significant cerebrovascular disease within 24 weeks of screening
* preexisting demyelinating disorder such as multiple sclerosis, or other severe neurological disorder
* major surgery within 4 weeks of screening, or scheduled to occur during the study, excluding diagnostic surgery
* previous treatment with total lymphoid irradiation
* history of any lymphoproliferative disorder such as Epstein Barr Virus, history of lymphoma, leukemia, or symptoms of current lymphatic or lymphoid disease
* Clinically significant depression, suicidal ideation, or previous history of suicidal behaviors
* Other medical or laboratory abnormality that may increase the risk of study participation
* Previous administration with an investigational product (drug or vaccine) within 30 days or of the first dose of study medicine
* Current use or incomplete appropriate washout period of any prohibited medication(s) or known exposure to anti-interferon beta (PF-06823859) or any type of anti-interferon beta therapy
* Prior SOC medication that does not fulfill the criteria
* Certain laboratory results from screening assessments that may interfere with study participation.
* Investigator site staff directly involved in the conduct of the study and their family members, site staff and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2027-07-28 (Estimated); Study Completion 2027-07-28 (Estimated)

PRIMARY OUTCOMES:
Moderate change in Total Improvement Score (TIS) | 24 weeks outside of the United States (US) and 52 weeks in the US
  Total Improvement Score 0 to 100 with higher scores indicating a better outcome.

SECONDARY OUTCOMES:
Change from baseline in Manual Muscle Testing - 8 designated muscles (MMT-8) | 24 weeks outside of the US and 52 weeks in the US
  Manual Muscle Testing (8 designated muscles) 0 to 150 with higher scores indicating a better outcome
Change from baseline in Cutaneous Dermatomyositis Disease Area and Severity Index Activity Score (CDASI-A) in participants with dermatomyositis (DM) | Week 24 outside the US
  Cutaneous Dermatomyositis Disease Area and Severity Index Activity Score 0 to 100 with higher scores indicating a worse outcome. Only participants with baseline CDASI-A score ≥14 will be assessed.
Change from baseline in Investigator Global Assessment severity scale (IGA) in participants with dermatomyositis | 24 and 52 weeks in the US only
  Investigator Global Assessment severity scale 0 to 4 with higher scores indicating a worse outcome. Only participants with baseline IGA ≥2 will be assessed
Corticosteroid (CS) dose assessment | 52 weeks
  Normalized Area Under the Curve (AUC) of corticosteroid dose
Moderate change in Total Improvement Score | 24 weeks in the US and 52 weeks outside of the US
  Total Improvement Score 0 to 100 with higher scores indicating a better outcome.
Change from baseline in Patient-Reported Outcomes Measurement Information System - Physical Function (PROMIS-PF) | 24 weeks outside of the US and 52 weeks in the US
  Patient-Reported Outcomes Measurement Information System - Physical Function 0 to 100 with higher scores indicating a better outcome
Change from baseline in 5-D Itch Scale Score | 24 weeks outside of the US and 52 weeks in the US
  5-D Pruritis Scale 5 to 25 with higher scores indicating a worse outcome. Only participants with baseline CDASI-A score ≥14 will be assessed.
Change from baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | 24 weeks outside of the US and 52 weeks in the US
  Functional Assessment of Chronic Illness Therapy - Fatigue 0 to 52 with higher scores indicating a better outcome
Response in corticosteroid tapering | 52 weeks US only
  At least 50% reduction from baseline or reduction in corticosteroid (CS) dose to <7.5 mg/day at Week 52 for participants with baseline CS dose ≥10 mg/day.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (124):
- United States (42):
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Glendale, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Glendale, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic in Arizona - Scottsdale, Scottsdale, Arizona
  - 200 UCLA Medical Plaza, Los Angeles, California
  - UCLA Clinical & Translational Research Center (CTRC), Los Angeles, California
  - UCLA, Los Angeles, California
  - Center for Clinical Research - Chapman Pavilion, Orange, California
  - UCI Douglas Hospital, Orange, California
  - UCI Health Center for Innovative Health Therapies, Orange, California
  - University of California - Irvine, Orange, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Lal Bhagchandani, M.D, Margate, Florida
  - University of Miami, Miami, Florida
  - University of Miami Dermatology Clinical Trials Unit, Miami, Florida
  - Unviversity of Miami, Miami, Florida
  - Omega Research Orlando, Orlando, Florida
  - IRIS Research and Development, LLC, Plantation, Florida
  - West Broward Pulmonary Consultants, Plantation, Florida
  - West Broward Rheumatology Associates, Tamarac, Florida
  - KU Clinical Research Center - Clinical and Translational Science Unit (CTSU), Fairway, Kansas
  - KU Clinical Research Center - Clinical and Translational Science Unit (CTSU) Rainbow, Kansas City, Kansas
  - University of Kansas Medical Center - Hoglund Brain Imaging Center, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - CTC - Brigham & Women's Hospital, Boston, Massachusetts
  - CTH - Brigham & Women's Hospital, Boston, Massachusetts
  - Washington University Pulmonary Function Laboratory, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Joseph S. and Diane H. Steinberg Ambulatory Care Center, Brooklyn, New York
  - NYU Langone Health - Clinical and Translational Science Institute Research Pharmacy, New York, New York
  - NYU Langone Health Clinical Research Center, New York, New York
  - NYU Langone Health, New York, New York
  - NYU Langone Radiology, New York, New York
  - NYU Langone Rusk Pulmonary Function Lab, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Arthritis & Rheumatology Research Institute, PLLC, Allen, Texas
  - Integrative Rheumatology of South Texas, Edinburg, Texas
  - Integrative Rheumatology of South Texas - Harlingen, Harlingen, Texas
  - Nerve & Muscle Center of Texas, Houston, Texas
  - Pulmonary and Sleep Center of the Valley, Weslaco, Texas
  - Rheumatology & Pulmonary Clinic, Beckley, West Virginia
- Argentina (5):
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Buenos Aires
  - CER medical Institute, Quilmes, Buenos Aires F.D.
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman, Tucumán Province
  - Hospital J. M. Ramos Mejía, Buenos Aires
  - Instituto de Reumatología, Mendoza
- UZ Leuven, Leuven, Vlaams-brabant, Belgium
- Bulgaria (2):
  - Medical Center Artmed, Plovdiv
  - Diagnostic Consultative Centre (DCC) - Foкus 5, Sofia
- China (15):
  - Anhui Provincial Hospital, Hefei, Anhui
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The first Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- France (2):
  - Centre Hospitalier Universitaire de Reims - l'Hôpital Maison Blanche, Reims
  - Hopitaux Universitaires de Strasbourg, Nouvel Hopital Civil, Strasbourg
- Germany (2):
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - Ludwig Maximilians University Munich Klinikum, München
- Debreceni Egyetem Klinikai Kozpont, Debrecen, Hungary
- India (3):
  - Medanta-The Medicity, Gurugram (Gurgaon), Haryana
  - CHARM HEALTHCARE PRIVATE LIMITED (Previously Dr Shenoy's Care Private Limited), Kochi, Kerala
  - Institute of Post Graduate Medical Education and Research and Seth Sukhlal Karnani Memorial Hospital, Kolkata, West Bengal
- Israel (3):
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Sourasky Medical Center, Tel Aviv, TELL ABĪB
- Italy (5):
  - IRCCS Istituto Clinico Humanitas, Rozzano, Milano
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM
  - Azienda Ospedaliero Universitaria Policlinico G.Rodolico-San Marco Di Catania, Catania
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Irccs Ospedale San Raffaele, Milan
- Japan (9):
  - Hospital of the university of occupational and environmental health, Kitakyushu-shi, Fukuoka
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Okayama City General Medical Center Okayama City Hospital, Okayama, Okayama-ken
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano, Osaka
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Institute of Science Tokyo Hospital, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
- Mexico (5):
  - Boca Clinical Trials Mexico S.C., Guadajalara, Jalisco
  - Centro Integral en Reumatologia, Guadalajara, Jalisco
  - Cryptex Investigación Clínica S.A. de C.V., Cuauhtémoc, Mexico City
  - CITER Centro de Investigación y Tratamiento de las Enfermedades Reumáticas, Mexico City, Mexico City
  - Private Practice - Dr. Miguel Cortes, Cuernavaca, Morelos
- Poland (10):
  - Pracownia Radiologiczna WIDOK-MED, Krakow, Lesser Poland Voivodeship
  - Małopolskie Centrum Kliniczne, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Plejady, Krakow, Lesser Poland Voivodeship
  - Lux Med, Krakow, Lesser Poland Voivodeship
  - 5 Wojskowy Szpital Kliniczny z Polikliniką SPZOZ, Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji, Warsaw, Masovian Voivodeship
  - Centrum Medycyny Oddechowej Robert Mroz spolka jawna, Bialystok, Podlaskie Voivodeship
  - INTER CLINIC Piotr Adrian Klimiuk, Bialystok, Podlaskie Voivodeship
  - Zaklad Diagnostyki Obrazowej HEM s.c., Bialystok, Podlaskie Voivodeship
  - Nova Reuma Domyslawska i Rusilowicz Spolka Partnerska Lekarza Reumatologa i Fizjoterapeuty, Bialystok, Podlaskie Voivodeship
- Narodny ustav reumatickych chorob, Piešťany, Slovakia
- South Korea (3):
  - Chonnam National University Bitgoeul Hospital, Gwangju, Kwangju-kwangyokshi
  - Kyung Hee University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Seoul National University Hospital, Seoul
- Spain (3):
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa CRUZ DE Tenerife
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Karolinska University Hospital Solna, Stockholm, Sweden
- Taiwan (6):
  - Chi Mei Medical Center, Tainan, Tainan
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (3):
  - Ankara University Ibni Sina Hospital, Ankara
  - Hacettepe Universite Hastaneleri, Ankara
  - Memorial Ankara Hastanesi, Ankara
- United Kingdom (2):
  - Queen Elizabeth University Hospital, Glasgow, Glasgow CITY
  - Salford Royal Hospital, Salford, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0251006